CLINICAL TRIAL: NCT03176264
Title: ElevatION: CRC-101: A Phase Ib Study of PDR001 in Combination With Bevacizumab and mFOLFOX6 as First Line Therapy in Patients With Metastatic MSS Colorectal Cancer
Brief Title: PDR001 in Combination With Bevacizumab and mFOLFOX6 as First Line Therapy in Patients With Metastatic MSS Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to company decision.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001I2101; 2017-000520-96 (EudraCT Number)
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: PDR001; immunotherapy; bevacizumab; mFOLFOX6; CRC; MMS; CMS4; ElevatION;CRC-101
MeSH Terms: conditions — Colorectal Neoplasms | interventions — spartalizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Phase Ib study, safety run-in (N=~6 pts) followed with an expansion (N=~86 pts). One single arm: PDR001 in combination with bevacizumab and mFOLFOX6
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental)
  Interventions: Drug: PDR001; Drug: bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: PDR001 — 400 mg every 4 weeks
Drug: bevacizumab — 5 mg/kg every 2 weeks
Drug: mFOLFOX6 — Combination of chemotherapy administered every 2 weeks: oxaliplatin (85mg/m2), 5-Fluorouracil (2400mg/m2) and folinic acid (=leucovorin, 400mg/m2)

SUMMARY:
This was a phase Ib study of PDR001 in combination with bevacizumab and mFOLFOX6 as first line therapy in patients with metastatic microsatellite stable (MSS) colorectal cancer. The study was to have assessed primarily, the safety and tolerability and then the efficacy of PDR001 in combination with bevacizumab and mFOLFOX6. Particular attention would have been paid to the level of activity of study drug combinations in CMS4 patients (retrospective analysis).

The study was terminated early due to company decision.

ELIGIBILITY:
Key inclusion criteria:

1. Patients with metastatic MSS colorectal adenocarcinoma.Note: MSI status will be performed locally by an immunohistochemistry (IHC) or PCR based test for eligibility.
2. Patients must provide a newly obtained or an archival tumor sample corresponding to CRC diagnosis (primary tumor) with sufficient tissue quality (qualified) for analysis (mandatory)
3. Patients must provide a newly obtained tumor tissue sample from a metastatic site (mandatory)
4. Patients who are naïve to systemic treatment in metastatic setting. Patients with previous neoadjuvant or adjuvant chemotherapy (that may have included oxaliplatin or investigational VEGF inhibitors) are eligible if the treatment was completed > 12 months before inclusion.
5. Patients with the presence of at least one lesion with measurable disease as per RECIST 1.1 guidelines. Lesions in previously irradiated areas should not be considered measurable unless they have clearly progressed since the radiotherapy.

9. Patients have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Key exclusion criteria:

1. Patients with MSI-H colorectal adenocarcinoma as defined per local assessment using standard of care testing
2. Patients with metastatic disease amenable to be resected with potentially curative surgery
3. Patients who have received any systemic treatment for metastatic disease.
4. Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PDL2, anti-CTLA-4 antibodies, other checkpoint inhibitors
5. Patients who had received radiation within 14 days prior to the first dose of study drug

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicity (DLT) | 12 months
Overall Response Rate (ORR) per investigator assessment using RECIST v1.1 | 19 months
  RECIST v1.1 = Response Evaluation Criteria in Solid Tumors v1.1

SECONDARY OUTCOMES:
Overall response rate (ORR) per central assessment using RECIST v1.1 | Baseline, every 8 weeks until progression per central assessment up to 1 year after last patient last visit
Overall survival (OS) | Every 3 months after last visit up to 1 year after last patient last visit
Progression free survival | Baseline, every 8 weeks until progression per central assessment up to 1 year after last patient last visit
Duration of response (DOR) | Baseline, every 8 weeks until progression per central assessment up to 1 year after last patient last visit
Disease control rate (DCR) | Baseline, every 8 weeks until progression per central assessment up to 1 year after last patient last visit
Time to response (TTR) | Baseline, every 8 weeks until progression per central assessment up to 1 year after last patient last visit
Ctrough | Through end of treatment completion, an average of 14 months
Cmax | Through end of treatment completion, an average of 14 months
Area under the curve (AUC) | Through end of treatment completion, an average of 14 months
Antidrug antibodies (ADA) | Through end of treatment completion, an average of 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17317
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=651